CLINICAL TRIAL: NCT04075773
Title: Brief Religious Alcohol Intervention
Acronym: BRAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Mary M. Tomkins, Graduate Research Assistant, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001734
Record Dates: First submitted 2019-08-28; First posted 2019-09-03 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Heavy Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either an intervention condition, where they will write about how their drinking relates to their religious identity, or to a control condition, where they will write about how their drinking relates to their age.
Who Masked: Participant, Care Provider
Masking Description: Participants will not be made aware of the purpose of the study. Research assistants, who interact with the participants, will not be made aware of which writing prompt any given participant will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Religious Prompt (Experimental): Participants will be provided a writing prompt that describes their self-reported drinking, then asks them to write for 5 to 10 minutes about how that drinking is associated with their self-reported religious identity. After completing that writing assignment, participants will be shown their response, and asked to spend 5 to 10 minutes describing how their drinking behaviors in the next month might change.
  Interventions: Behavioral: Expressive Writing
- Age Prompt (Sham Comparator): Participants will be provided a writing prompt that describes their self-reported drinking, then asks them to write for 5 to 10 minutes about how that drinking is associated with their self-reported age. After completing that writing assignment, participants will be shown their response, and asked to spend 5 to 10 minutes describing how their drinking behaviors in the next month might change.
  Interventions: Behavioral: Expressive Writing

INTERVENTIONS:
Behavioral: Expressive Writing — The participants are asked to write for a period of time about specific concepts so that they think carefully and cognitively process the information they are generating.

SUMMARY:
This study is a trial of a brief alcohol intervention, a brief expressive writing intervention that incorporates religious identity.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 29 years old
* Have had a binge episode (4/5 drinks on one occasion for women/men) at least once in the past month
* UH students

Exclusion Criteria:

* Participants who are currently enrolled in treatment for alcohol or other substances
* Participants who have been diagnosed with and/or treated for verbal learning disabilities

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Change in the Timeline Follow-Back one month following the intervention | It will be assessed before the intervention and one month following the intervention.
  Participants report number of drinks consumed each day over the last month.

SECONDARY OUTCOMES:
Chang in the Young Adult Alcohol Consequences Questionnaire one month following the intervention | It will be assessed before the intervention and one month following the intervention.
  Participants respond to a list of common consequences of alcohol use indicating whether or not they have experienced them. The scale name is the "Young Adult Alcohol Consequences Questionnaire" (Read, Kahler, Strong, & Colder, 2006). The construct of interest measured by this scale is the alcohol problems experienced by the participant. The total score is used, and the range for the total score is 0 to 48.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Tomkins, M.S., Principal Investigator — University of Houston
Locations (1):
- University of Houston Psychology Department, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not have any plans at this time to share individual participant data with other researchers.